CLINICAL TRIAL: NCT04659954
Title: Feasibility and Acceptability Study of the "O'Dide" Application in People Suffering From an Addiction
Acronym: FA-O'DIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut de Recherche en Santé Publique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/20/0367
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Substance-Related Disorders; Personality Disorders
Keywords: E health; Application; Substance use disorders; Personality disorders; Care observance
MeSH Terms: conditions — Substance-Related Disorders; Personality Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Application O'DIDE (Experimental): The subjects will use the application O'DIDE during 8 weeks
  Interventions: Other: Application O'DIDE

INTERVENTIONS:
Other: Application O'DIDE — The intervention is the use of an application that aimed to favorize contact between the patient and the care team between the consultations.

SUMMARY:
Substance Use Disorders (SUD) are associated with cognitive schemas that lead to care attrition and mistrust towards care. Considering this within SUD management, it is important to establish a confident relation between the patient and the care team to favorize acre observance. However, it demands an important availability of the healthcare team, allowing for frequent interactions at all times, including at night and during days off. With the present study, the investigator postulated that an application called Ô DIDE for Digital Interaction for Detoxification Engagement, that aims to help the caregivers maintaining a link with the patient in order to facilitate confidence in the relationship, could favorize care observance especially consumption report.

DETAILED DESCRIPTION:
The present research aims to assess the feasibility of the "Ô DIDE" application after 8 weeks of use by patients treated for a disorder related to substance use at the Toulouse University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Suffering from any type of addiction, with an active addiction requiring weekly monitoring of consumption
* Possessing an Android smartphone or having access to an Android smartphone and having access to an internet connection
* Able to read and understand French
* Affiliated or beneficiary of a social security scheme.
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patient with cognitive or psychiatric disorders that may affect their ability to consent
* Participation in another protocol involving a modification of the treatment for addiction
* Person under legal protection, guardianship or curatorship
* Known or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of use of the application O'DIDE during 8 weeks | 8 weeks
  Percentage of patients who logged on at least once a week to the application during the 8 weeks of availability of the O'DIDE application

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Salles, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University hospital of Toulouse, Toulouse, France

REFERENCES:
- [Derived] Stocker A, Navarro N, Schmitt L, Delagnes M, Doualle A, Mallard V, Entajan F, Guivarc'h K, Masse P, Chaigneau L, Bonneau B, Lapeyre-Mestre M, Arbus C, Yrondi A, Salles J. Acceptability of "DIDE", a mobile application designed at facilitating care adherence of patients with substance use disorder. Addict Sci Clin Pract. 2024 Oct 15;19(1):72. doi: 10.1186/s13722-024-00500-7. PMID 39407238